CLINICAL TRIAL: NCT02600780
Title: Febuxostat (Zurig) Efficacy & Safety Trial in Comparison With Allopurinol in Hyperuricemic Subjects With or Without Gout
Brief Title: Zurig (Febuxostat) 40mg Efficacy and Safety Trial
Acronym: ZEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUHS-GTZ-MD-001-13
Record Dates: First submitted 2015-11-02; First posted 2015-11-09 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Hyperuricemia
Keywords: Febuxostat; Efficacy; Safety; Allopurinol; Hyperuricemia; Zurig; Getz Pharma
MeSH Terms: conditions — Hyperuricemia | interventions — Febuxostat; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allopurinol (Active Comparator): Allopurinol 300mg Tablets once daily for 90 days
  Interventions: Drug: Allopurinol
- Febuxostat (Experimental): Febuxostat 40mg Tablets once daily for 90 days
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — Comparison of two anti-hyperuricemic molecules
  Other Names: Zurig
  Arms: Febuxostat
Drug: Allopurinol — Comparison of two anti-hyperuricemic molecules
  Arms: Allopurinol

SUMMARY:
Febuxostat is a potent, nonpurine, selective inhibitor of Xanthine oxidase that exhibits antihyperuricemic activity by reducing the formation of uric acid. The investigators conducted an interventional, two-arm, randomized, open label pilot study on patients with serum urate level ≥ 6.8 mg/dL. Patients were treated with Febuxostat 40 mg Tablets or Allopurinol 300 mg Tablets once daily dose for 90 days to determine the efficacy and safety of Febuxostat in comparison with Allopurinol in Hyperuricemic Subjects with or without Gout.

DETAILED DESCRIPTION:
Patients with hyperuricemia (with or without Gout) were randomized into two groups. One was treated with Febuxostat 40 mg Tablets and other with Allopurinol 300 mg Tablets once daily for 3 months period.

Gender, age, height, weight, creatinine and ALT levels, co-morbidities and other complications were monitored at screening and as per eligibility criteria 50 patients were enrolled in the study. Efficacy was determined by monitoring serum uric acid levels during and at the end of treatment. The safety profile has also been monitored during the treatment period. Investigator collected and recorded all the data of visits in CRF which was analyzed through SPSS version 20.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders from 18 to 75 years of age
2. Must have a serum urate level ≥ 6.8 milligram per deciliter (mg/dL) and/or subjects recruited with Gout; must meet American College of Rheumatology criteria for Gout.
3. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
4. Patient willingly provides written informed consent

Exclusion Criteria:

1. History of significant concomitant illness
2. Active liver disease (SGPT> 1.5 times the upper limit of normal range)
3. Severe renal impairment (Serum Creatinine level >2mg/dl)
4. Any other significant medical condition that would interfere with the treatment, safety or compliance with the protocol, as defined by the investigator
5. Cardiac disease or stroke (current or previous history)
6. Has a known history of infection with hepatitis B, hepatitis C, or HIV
7. Has a history of cancer within 5 years prior to the first dose of study medication
8. Has a known hypersensitivity to febuxostat or allopurinol or any components of their formulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Serum uric acid levels | 3 months
  To determine the efficacy of Febuxostat once daily with Allopurinol once daily in hyperuricemic subjects for 3 months

SECONDARY OUTCOMES:
Safety Assessment: number of participant with adverse events | At week 2, week 4 and week 12
  To determine the number of patients treated with Febuxostat once daily with Allopurinol once daily who experience any adverse drug reaction. All ADR are reported as per patient information leaflet

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Mahmood, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Krishnan E, Svendsen K, Neaton JD, Grandits G, Kuller LH; MRFIT Research Group. Long-term cardiovascular mortality among middle-aged men with gout. Arch Intern Med. 2008 May 26;168(10):1104-10. doi: 10.1001/archinte.168.10.1104. PMID 18504339
- [Background] Khanna D, Fitzgerald JD, Khanna PP, Bae S, Singh MK, Neogi T, Pillinger MH, Merill J, Lee S, Prakash S, Kaldas M, Gogia M, Perez-Ruiz F, Taylor W, Liote F, Choi H, Singh JA, Dalbeth N, Kaplan S, Niyyar V, Jones D, Yarows SA, Roessler B, Kerr G, King C, Levy G, Furst DE, Edwards NL, Mandell B, Schumacher HR, Robbins M, Wenger N, Terkeltaub R; American College of Rheumatology. 2012 American College of Rheumatology guidelines for management of gout. Part 1: systematic nonpharmacologic and pharmacologic therapeutic approaches to hyperuricemia. Arthritis Care Res (Hoboken). 2012 Oct;64(10):1431-46. doi: 10.1002/acr.21772. No abstract available. PMID 23024028
- [Result] Becker MA, Chohan S. We can make gout management more successful now. Curr Opin Rheumatol. 2008 Mar;20(2):167-72. doi: 10.1097/BOR.0b013e3282f54d03. PMID 18349746
- [Result] Okamoto K, Eger BT, Nishino T, Kondo S, Pai EF, Nishino T. An extremely potent inhibitor of xanthine oxidoreductase. Crystal structure of the enzyme-inhibitor complex and mechanism of inhibition. J Biol Chem. 2003 Jan 17;278(3):1848-55. doi: 10.1074/jbc.M208307200. Epub 2002 Nov 5. PMID 12421831
- [Result] Takano Y, Hase-Aoki K, Horiuchi H, Zhao L, Kasahara Y, Kondo S, Becker MA. Selectivity of febuxostat, a novel non-purine inhibitor of xanthine oxidase/xanthine dehydrogenase. Life Sci. 2005 Mar 4;76(16):1835-47. doi: 10.1016/j.lfs.2004.10.031. Epub 2005 Jan 18. PMID 15698861